CLINICAL TRIAL: NCT06222892
Title: A Phase 1, Open-label Study to Investigate the Pharmacokinetics and Safety of Camlipixant in Male and Female Participants Aged 18-75 Years of Age With Hepatic Impairment Compared to Matched Healthy Participants With Normal Hepatic Function
Brief Title: A Study of Camlipixant in Male and Female Healthy Participants and Participants With Hepatic Impairment Aged 18-75 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221852
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Cough
Keywords: Camlipixant; Healthy participants; Hepatic Impairment; Pharmacokinetic; Safety
MeSH Terms: conditions — Cough

STUDY DESIGN:
Masking Description: This will be an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Moderate HI Participants (Experimental): Participants with moderate HI received a single dose of camlipixant 50 milligrams (mg) tablet orally on Day 1 in the fasted state.
  Interventions: Drug: Camlipixant
- Part 1: Matched Healthy Participants to Moderate HI (Experimental): Healthy participants (matched to participants with moderate HI) received a single dose of camlipixant 50 mg tablet orally on Day 1 in the fasted state.
  Interventions: Drug: Camlipixant
- Part 2: Severe HI Participants (Experimental): Participants with severe HI received a single dose of camlipixant 50 mg tablet orally on Day 1 in the fasted state.
  Interventions: Drug: Camlipixant
- Part 2: Matched Healthy Participants to Severe HI (Experimental): Healthy participants (matched to participants with severe HI) received a single dose of camlipixant 50 mg tablet orally on Day 1 in the fasted state.
  Interventions: Drug: Camlipixant

INTERVENTIONS:
Drug: Camlipixant — Camlipixant was administered.

SUMMARY:
The purpose of this study is to assess the effect of Hepatic impairment (HI) on the Pharmacokinetic (PK) profile and safety of Camlipixant.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all participants

* Adult male or female participant, greater than or equals to (>=) 18 years and less than or equals to (<=) 75 years of age at the screening visit.
* Male and female participants must follow protocol-specified contraception guidance.

Guidance for Female Participants

a. Female participants of childbearing potential must agree to one of the following methods of contraception: i. Hysteroscopic sterilization or bilateral tubal ligation at least 6 months prior to dosing.

ii. Non-hormonal releasing intrauterine device (IUD) or hormonal contraceptives (e.g., oral, IUD, vaginal ring, transdermal patch, depot, implantable, etc.) for at least 3 months prior to dosing and with either a physical (e.g., condom, diaphragm, or other) or a chemical (e.g., spermicide) barrier method from the time of the screening visit.

b. In addition, female participants of childbearing potential will be advised to keep the same birth control method for at least 30 days after dosing.

c. Female participant must agree not to donate ova from dosing until at least 30 days after dosing.

Guidance for male participants. a. Male participants who are not vasectomized for at least 4 months prior to dosing and who are sexually active with a female partner of childbearing potential must be willing to use one of the following acceptable contraceptive methods from dosing until 90 days after dosing.

i. Simultaneous use of condom and hormonal contraceptive (e.g., oral, IUD, vaginal ring, patch, depot, implantable, etc.) or non-hormonal intrauterine device used for at least 3 months prior to dosing for the female partner.

ii. Simultaneous use of condom and a diaphragm or cervical cap with spermicide for the female partner.

b. No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to dosing. A male who has been vasectomized less than 4 months prior to dosing must follow the same restrictions as a non-vasectomized male.

1. Female Participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: Is a woman of non-childbearing potential (WONCBP) OR Is a Woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, with a failure rate of <1 percent (%), during the study intervention period and for at least 14 days after the last dose of study intervention. The investigator should evaluate potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of study intervention.
2. A WOCBP must have a negative highly sensitive pregnancy test urine or serum as required by local regulations) within specify timeframe before the first dose of study intervention. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
3. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

   * Participants must weigh at least 50 kilogram (kg) and have a Body mass index (BMI) >= 18.0 and <= 40.0 kilograms per square meter (kg/m^2), at the screening visit.
   * Continuous non-smoker who has not used nicotine- and tobacco-containing products or light smoker (<= 5 cigarettes/day or the equivalent) for the last 3 months prior to study screening.
   * Participant who understands the study procedures in the informed consent form (ICF) and is willing and able to comply with the protocol.

Additional inclusion criteria for hepatic impaired participants.

* Participants aside from HI, be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, ECGs, and screening clinical laboratory profiles, as deemed by the Principal Investigator (PI) or designee, including the following:

  1. Seated blood pressure is >= 90/40 millimeters of mercury (mmHg) and <= 160/100 mmHg at the screening visit.
  2. Seated heart rate is >= 40 beats per minute (bpm) and <= 99 bpm at the screening visit.
  3. Corrected value of the interval between the Q and T waves on the electrocardiogram tracing, corrected QT interval using Fridericia formula (QTcF) is <= 480 milliseconds (msec) and has ECG findings considered normal or not clinically significant by the PI or designee at the screening visit.
  4. Estimated creatinine clearance >= 80 milliliters per minute (mL/min) at the screening visit.
  5. Total bilirubin <= 6 milligrams per deciliters (mg/dL).
* Has a score on the Child-Pugh scale at the screening visit as follows:

  a. Severe HI: >= 10 and <= 15; or Moderate HI: >= 7 and <= 9; or Mild HI: >= 5 and <= 6.
* Participant has stable HI as defined by a diagnosis of chronic (>= 6 months), stable (no acute episodes of illness within 30 days prior to dosing due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology.

Additional inclusion criteria for healthy control participants:

* Medically healthy participants with no clinically significant medical history, physical examination, screening clinical laboratory profiles, vital signs and ECGs, as deemed by the PI or designee, including the following:

  1. Seated blood pressure is >= 90/40 mmHg and <= 140/90 mmHg at the screening visit.
  2. Seated heart rate is >= 40 bpm and <= 99 bpm at the screening visit.
  3. QTcF interval is <= 450 msec and has ECG findings considered normal or not clinically significant by the PI or designee at the screening visit.
  4. QTc <= 480 msec in participants with bundle branch block.
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), direct bilirubin, indirect bilirubin, and total bilirubin within normal ranges at the screening visit and check-in. Only abnormal values up to 1.5 times upper limit of normal may be repeated once.

Exclusion Criteria:

Exclusion criteria for all participants:

* Mentally or legally incapacitated participants or has significant emotional problems at the time of the screening visit or are expected during the conduct of the study.
* Participants with surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the participant's safety in case of participation in the study.
* Participants with history or presence of liver or other solid organ transplant.
* Participants with history of acute pancreatitis within 1 year of study entry.
* Participant with history or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
* Participant who has received any Coronavirus Disease-2019 (COVID-19) vaccine within 14 days prior to dosing.
* Participant who is unable to refrain from or anticipates the use of prohibited prescription or non-prescription medication, herbal remedies, or supplements.
* Participant with history or presence of drug abuse within the past 6 months prior to dosing. Positive drug screen due to prescription drug use in hepatic impaired participants will be allowed if approved by PI on a case by case basis.
* Participation in another clinical study within 30 days (or 5 half-lives, whichever is longer) prior to dosing. The 30 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.
* Participants with positive pre-study drug/alcohol screen, including tetrahydrocannabinol (THC) at the screening visit or at check-in, unless the positive drug test is due to prescription drug use that is approved by the PI or designee and sponsor.
* Participants with positive results for Human immunodeficiency virus (HIV).
* Participants has positive coronavirus Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) rapid test and/or positive polymerase chain reaction test (based on local procedures) at check-in.
* Participants with presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study intervention.
* Participants with positive hepatitis C antibody test result at screening or within 3 months prior to starting study intervention.
* Participants with unhealthy alcohol use, defined as use more than 24 grams (g) pure alcohol per day for male and 12 g for female (12 g equals to approximately 300 milliliters [mL] beer, 100 mL wine, or 25 mL spirits).
* Participant has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 30 days prior to dosing.
* Donation of blood or plasma greater than 400 mL within the last 90 days prior to dosing.
* Donation of bone marrow within the last 6 months prior to dosing.

Additional exclusion criteria for hepatic impaired participants:

* Participant with history or presence of clinically significant medical or psychiatric condition or disease (aside from HI) in the opinion of the PI or designee and Sponsor medical representative.

Additional exclusion criteria for healthy control participants:

* Participant with history or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee and Sponsor medical representative.
* Participant with history or presence of alcoholism or drug abuse within the past 2 years prior to dosing.
* Female participant with a positive pregnancy test at the screening visit or at check-in or who is lactating (also applies to female HI participants).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 2 parts - Part 1 and Part 2. In Part 1, participants with moderate hepatic impairment (HI) and matched healthy participants were enrolled. Based on the pharmacokinetic (PK) and safety data from Part 1, only participants with severe HI and their matched healthy participants were enrolled in Part 2, while participants with mild HI were not enrolled.
Pre-assignment Details: A total of 32 participants (16 in Part 1 and 16 in Part 2) were enrolled in this study.
Period: Part 1 (Up to 17 Days)
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2 (Up to 17 Days)
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Started | 0 | 0 | 8 | 8
Completed | 0 | 0 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Moderate HI Participants: Participants with moderate HI received a single dose of camlipixant 50 mg tablet orally on Day 1 in the fasted state.
- Total: Total of all reporting groups
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 58.8 (9.92) | 56.8 (6.96) | 49.9 (9.95) | 51.6 (9.32) | 54.3 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 2 | 12
  Male | 4 | 4 | 6 | 6 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC[0-inf]) of Camlipixant
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of camlipixant. PK analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: The analysis was performed on the PK Analysis Set that included all participants who received study intervention and who had at least 1 non-missing PK assessment (non-quantifiable [NQ] values were considered as non-missing values).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Hours*nanograms per milliliter | 5811 (22.7) | 4735 (19.0)

2. Primary Outcome: Part 2: AUC(0-inf) of Camlipixant
Description: Blood samples were collected at indicated time points for PK analysis of camlipixant. PK analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: The analysis was performed on the PK Analysis Set that included all participants who received study intervention and who had at least 1 non-missing PK assessment (NQ values were considered as non-missing values).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Hours*nanograms per milliliter | 7827 (39.9) | 4662 (46.9)

3. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Nanograms per milliliter | 1317 (33.5) | 960.0 (30.7)

4. Primary Outcome: Part 2: Cmax of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Nanograms per milliliter | 1228 (38.9) | 985.8 (29.8)

5. Secondary Outcome: Part 1: Number of Participants With Any Adverse Event (AE), Serious Adverse Event (SAE), and Adverse Event of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAEs are defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in a participant's offspring; abnormal pregnancy outcomes; is a suspected transmission of any infectious agent via an authorized medicinal product; or other situations as per medical and scientific judgement of the Investigator. AESIs are AEs of scientific interest specific to the drug class. AESIs for this study include the following but not limited to taste disturbance (dysgeusia, hypogeusia, ageusia), oral paresthesia and oral hypoesthesia. Number of participants with any AE, SAE, or AESI were reported.
Time Frame: Up to 17 days
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Participants
  Any AE | 0 | 0
  Any SAE | 0 | 0
  Any AESI | 0 | 0

6. Secondary Outcome: Part 2: Number of Participants With Any AE, SAE, and AESI
Description: as for outcome 5
Time Frame: Up to 17 days
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Participants
  Any AE | 2 | 0
  Any SAE | 0 | 0
  Any AESI | 0 | 0

7. Secondary Outcome: Part 1: Number of Participants With Clinically Significant Changes in Clinical Chemistry Parameters
Description: Blood samples were collected to analyze clinical chemical parameters: blood urea nitrogen (BUN)/urea, potassium, creatinine, sodium, calcium, glucose [fasting/non-fasting], creatine phosphokinase (CPK), serum albumin concentration, serum alpha-1-glycoprotein concentration, aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT), alkaline phosphatase, total bilirubin, direct bilirubin, indirect bilirubin and total protein. Number of participants with clinically significant changes in clinical chemistry parameters has been reported. Clinical significance was determined by the Investigator.
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

8. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Changes in Clinical Chemistry Parameters
Description: Blood samples were collected to analyze clinical chemical parameters: BUN/urea, potassium, creatinine, sodium, calcium, glucose [fasting/non-fasting], CPK, serum albumin concentration, serum alpha-1-glycoprotein concentration, AST/SGOT, ALT/SGPT, alkaline phosphatase, total bilirubin, direct bilirubin, indirect bilirubin and total protein. Number of participants with clinically significant changes in clinical chemistry parameters has been reported. Clinical significance was determined by the Investigator.
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

9. Secondary Outcome: Part 1: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples were collected to analyze hematology parameters: platelet count, red blood cell (RBC) count, RBC indices (mean corpuscular volume [MCV], mean corpuscular hemoglobin [MCH], percent reticulocytes), white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophil, basophils), hemoglobin, and hematocrit. Number of participants with clinically significant changes in hematology parameters has been reported. Clinical significance was determined by the Investigator.
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

10. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples were collected to analyze hematology parameters: platelet count, RBC count, RBC indices (MCV, MCH, percent reticulocytes), WBC count with differential (neutrophils, lymphocytes, monocytes, eosinophil, basophils), hemoglobin, and hematocrit. Number of participants with clinically significant changes in hematology parameters has been reported. Clinical significance was determined by the Investigator.
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

11. Secondary Outcome: Part 1: Number of Participants With Clinically Significant Changes in Urinalysis
Description: Urine samples were collected to analyze urinalysis parameters: specific gravity; and potential of hydrogen (pH), glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase which were analyzed by dipstick. Number of participants with clinically significant changes in urinalysis parameters has been reported. Clinical significance was determined by the Investigator.
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

12. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Changes in Urinalysis
Description: Urine samples were collected to analyze urinalysis parameters: specific gravity; and pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase which were analyzed by dipstick. Number of participants with clinically significant changes in urinalysis parameters has been reported. Clinical significance was determined by the Investigator.
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

13. Secondary Outcome: Part 1: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital signs including systolic and diastolic blood pressure, pulse rate, respiratory rate, and temperature were measured. Blood pressure and pulse rate measurements were performed with participants in a seated position for at least 5 minutes, except when they were supine or semi-reclined because of study procedures and/or AEs (such as nausea, dizziness). Number of participants with abnormal clinically significant changes in vital signs has been reported. Clinical significance was determined by the Investigator.
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

14. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Changes in Vital Signs
Description: as for outcome 13
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

15. Secondary Outcome: Part 1: Number of Participants With Clinically Significant Changes in 12 Lead Electrocardiogram (ECG) Findings
Description: ECG values included measurements of heart rate, PR interval, QRS interval, uncorrected QT interval, and corrected QT interval using Fridericia formula (QTcF). 12-lead ECG was recorded with the participant in a supine position for at least 5 minutes. Number of participants with clinically significant 12-lead ECG findings has been reported. Clinical significance was determined by the Investigator.
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

16. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Changes in 12 Lead ECG Findings
Description: ECG values included measurements of heart rate, PR interval, QRS interval, uncorrected QT interval, and QTcF. 12-lead ECG was recorded with the participant in a supine position for at least 5 minutes. Number of participants with clinically significant 12-lead ECG findings has been reported. Clinical significance was determined by the Investigator.
Time Frame: Up to Day 5
Population: The analysis was performed on the Safety Analysis Set that included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

17. Secondary Outcome: Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Hours | 0.750 [0.25 to 2.50] | 1.000 [0.50 to 2.50]

18. Secondary Outcome: Part 2: Tmax of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Hours | 0.750 [0.25 to 2.50] | 0.875 [0.47 to 2.50]

19. Secondary Outcome: Part 1: Terminal Elimination Half-life (T1/2) Following Administration of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Hours | 6.101 (46.8) | 5.809 (14.4)

20. Secondary Outcome: Part 2: T1/2 Following Administration of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Hours | 6.626 (17.1) | 7.855 (56.3)

21. Secondary Outcome: Part 1: Apparent Oral Clearance (CL/F) of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Liters per hour | 8.605 (22.7) | 10.56 (19.0)

22. Secondary Outcome: Part 2: CL/F of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Liters per hour | 6.388 (39.9) | 10.73 (46.9)

23. Secondary Outcome: Part 1: Apparent Oral Volume of Distribution (Vz/F) of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI
Number analyzed (Participants) | 8 | 8
Liters | 75.74 (36.3) | 88.49 (20.4)

24. Secondary Outcome: Part 2: Vz/F of Camlipixant
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
Number analyzed (Participants) | 8 | 8
Liters | 61.06 (32.5) | 121.6 (42.5)

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs, and non-SAEs were collected up to 17 days for both Part 1 and Part 2
Description: Safety Analysis Set included all participants who received study intervention.
Arm/Group | Part 1: Moderate HI Participants | Part 1: Matched Healthy Participants to Moderate HI | Part 2: Severe HI Participants | Part 2: Matched Healthy Participants to Severe HI
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 2/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Moderate HI Participants (N=8) | Part 1: Matched Healthy Participants to Moderate HI (N=8) | Part 2: Severe HI Participants (N=8) | Part 2: Matched Healthy Participants to Severe HI (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT06222892/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT06222892/SAP_001.pdf